CLINICAL TRIAL: NCT07182084
Title: Comparison of Proprioception and Manual Skills Between Physiotherapists and Other Healthcare Professionals
Brief Title: Proprioception and Manual Skills
Status: Not yet recruiting | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Associate Professor, Kahramanmaras Sutcu Imam University
Other Study IDs: Comparison of Proprioceptive
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Proprioception; Physiotherapist; Health Professionals

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/study group: Healthcare professionals(physiotherapist/nurse/midwife, doctor) living in Kahramanmaraş province

SUMMARY:
The proprioception refers to a person's awareness of the position, velocity, and weight of any body part in space. Proprioception consists of joint position sense and joint movement sense.Proprioception arises from the coordination of many different receptors, and it is assumed that these receptors are concentrated in muscles, tendons, joint capsules, and ligaments. Examples of proprioceptors include the golgi tendon organ, muscle spindles, pacinian corpuscles, and free nerve endings. Proprioceptive sense is closely related to many movements performed to perform daily activities. Proprioceptive sense is considered one of the most important resources in the development of task-specific neuroplasticity.The healthcare sector comprises individuals from many professional groups. Each professional group reaches professional competence by undergoing specific educational and training stages. Physiotherapists are one of these professional groups. To fulfill their professional duties, physiotherapists are expected to possess core competencies such as patient assessment using various manual methods, clinical decision-making, technical, communication, and therapeutic skills. Furthermore, a key difference distinguishing physiotherapists from other professions is their extensive manual contact with patients during assessment and treatment programs. Members of this professional group receive various training programs in manual therapy methods during their undergraduate studies. They undergo various qualifications that develop their manual skills and conduct assessment, treatment, and rehabilitation using various manual methods throughout their professional careers. The hand, with its complex structure, is one of the most prominent parts of the human body. Despite accounting for 0.6% of body weight and 2% of body surface area, the hand accounts for over 20% of the motor and sensory homunculus, demonstrating the importance and complexity of the hand's functional structure. The hand's ability to perform these complex skills depends not only on motor ability but also on two excellent sensory systems: proprioception and the sense of touch.It is thought that upper extremity proprioceptive sense and manual dexterity may vary among healthcare professionals. The literature primarily focuses on studies evaluating the proprioceptive sense and manual dexterity of dentists. However, it is noteworthy that studies have not compared the differences in proprioceptive sense and manual dexterity among healthcare professionals. Therefore, the purpose of this study was to compare proprioceptive sense and manual dexterity between physiotherapists and other healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are healthcare professionals (doctors, physiotherapists, nurses, and midwives)
* Individuals who have worked in the field for at least one year
* Individuals who have full range of motion in the upper extremity
* Individuals who speak and communicate in Turkish

Exclusion Criteria:

* - Individuals with any neurological problem (Parkinson's, hemiplegia, etc.)
* Individuals experiencing predominant upper extremity edema or pain due to musculoskeletal trauma in the last 6 months
* Pregnant individuals
* Blind individuals
* Individuals diagnosed with rheumatological diseases such as rheumatoid arthritis or osteoarthritis
* Individuals with sensory or motor loss in the upper extremity

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Doctors, physiotherapists, nurses and midwives who work in the Kahramanmaraş city center and agree to participate in the study will be included.
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Proprioception Measurement | on the first day of assessment
  All participants will undergo upper extremity (shoulder, elbow, wrist) proprioception assessment. Participants will complete a practice trial before each test. In the practice trial, target angles will be presented to the participant not verbally, but by positioning the joints for 5 seconds. After confirming that the participant has grasped the position with the "OK" command, the participant will return to the neutral position. A 5-second break will be allowed between repetitions, and the next joint range of motion will be performed when the participant is ready (30). Tests will be measured with a goniometer without contact, and absolute angular differences will be recorded. Each test will be performed twice on both extremities, and the average of absolute angular differences will be calculated. Dominant and non-dominant hands will be determined based on the answer to the question "Which hand do you write with?" Participants' eyes will be covered with an eye patch during the tests.
Purdue Pegboard Test (PPT) | on the first day of assessment
  The PPT consists of a board with two parallel rows of 25 holes into which cylindrical metal nails are inserted. The evaluator's guide contains the nail board, 25 pins, 45 washers, and 55 nails. Participants are asked to take a pin from a cup and insert it into one of the holes on the board, starting with the first hole closest to the cup. The objective is to fill as many holes as possible with nails within a 30-second time limit. The test is performed simultaneously with the dominant limb first, then the non-dominant limb, and finally both limbs. Scores are awarded based on the number of pins, washers, and nails.

SECONDARY OUTCOMES:
sosyodemographic form | in the first day of assesment
  Personal Information Form: Demographic information (age, height, weight, education level, dominant hand), frequency of upper extremity use outside of normal tasks (based on VAS), and whether or not the participant engages in tasks requiring fine manual dexterity will be questioned.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice adıgüzel tat, Associate Professor, Principal Investigator — Kahramanmaras Sutcu Imam University; abdulkadir ertürk, Msc, Principal Investigator — Kahramanmaras Sutcu Imam University; Yusuf Şinasi Kırmacı, Asisstant Prof, Study Chair — Kahramanmaras Sutcu Imam University; Tuğçe Simay Özbay, Msc, Study Chair — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaraş Sütçü imam University, Kahramanmaraş, Onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No